CLINICAL TRIAL: NCT01928680
Title: Phase II Study of Capecitabine and Cisplatin in Anthracycline and Taxanes-pretreated Metastatic Triple Negative Breast Cancer Patients
Brief Title: Phase II Study of Capecitabine and Cisplatin to Treat Metastatic Triple Negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Li Qiao, MD, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LQ0001; CAMS-LQ0001 (Other: cams)
Record Dates: First submitted 2013-05-01; First posted 2013-08-27 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Metastatic Breast Cancer
Keywords: Triple Negative Breast Cancer, Cisplatin, Capecitabine
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cisplatin/Capecitabine (Experimental): Capecitabine 1000mg/m2 orally Bid on day 1 to day 14 plus Cisplatin 75mg/m2 on day1 of each 21 day cycle, until progression or untolerable toxicity.
  This is a single arm phase II clinical trial.
  Interventions: Drug: Cisplatin/Capecitabine

INTERVENTIONS:
Drug: Cisplatin/Capecitabine — Cisplatin/Capecitabine: Capecitabine 1000mg/m2 orally Bid on day 1 to day 14 plus Cisplatin 75mg/m2 on day1 of each 21 day cycle, until progression or untolerable toxicity
  Other Names: Xeloda

SUMMARY:
It is a phase II trial to explore the efficacy and safety of cisplatin plus capecitabine in anthracycline and taxane-pretreated metastatic triple negative breast cancer patients.

DETAILED DESCRIPTION:
Cisplatin contained regimens have been demonstrated to be effective in metastatic triple negative breast cancer patients in some phase II clinical trials. Meanwhile, Capecitabine is also a highly effective choice for metastatic breast cancer with considerable duration of response. Combination of cisplatin and capecitabine have been proved effective in metastatic breast cancer in several phase II trials. This study is aimed to investigate the efficacy and safety of this combination in triple negative breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Written and signed informed consent prior to beginning specific protocol procedures.
* Pathologically confirmed Estrogen Receptor(ER), Progesterone Receptor(PR) and Human Epidermal growth factor Receptor HER-2) negative ("triple negative") breast cancer and documented metastatic or locally advanced disease.

Measurable disease - with at least 1 lesion measurable by radiological method

* KPS>=70
* 18 to 70 years old women
* Previously treated with an anthracycline and a taxane
* Hormone therapy for early-stage or metastatic breast cancer was permitted if hormonal receptor positive.
* Treatment with Herceptin for early-stage or metastatic breast cancer is permitted if HER2 positive
* Laboratory requirements:

  * Hematology Absolute neutrophil count>=1,500 /μl; Platelets>=100,000 /μl; Hemoglobin>=10 g/dl
  * Liver function Total bilirubin<=2 times ULN ASAT (SGOT) and ALAT (SGPT)<=2.5 times UNL without liver metastasis or <=5.0 times if liver metastasis Glucose<=200 mg/dL
  * Renal function Serum creatinine<=140 mol/l
* Life expectancy of at least 12 weeks
* Patients must be accessible for treatment and follow-up.
* Patients should have recovered from the acute reversible effects of prior treatment. This generally means at least 3 weeks should have elapsed since prior chemotherapy, adjuvant or Neoadjuvant treatment. and at least 4 weeks since prior (radical) radiotherapy or major surgery

Exclusion Criteria:

* Women who are pregnant or breast feeding
* History of brain and/or leptomeningeal metastases
* Past or current history of malignant neoplasm other than breast carcinoma, except for curatively treated non melanoma skin cancer, in situ carcinoma of the cervix or other cancer curatively treated and with no evidence of disease for at least 5 years
* Pre-existing neuropathy grade 1 according to the NCIC-CTC 3.0
* Psychiatric disorders or other conditions which would prevent pt. compliance
* Other serious illness or medical condition:
* Congestive heart failure, or unstable angina pectoris, previous history of myocardial infarction within 6 month prior to study entry, uncontrolled hypertension as determined by the Investigator or high risk uncontrolled, arrhythmia.
* History of significant neurological or psychiatric disorders including psychotic disorders, dementia of seizures that would prohibit the understanding and giving of informed consent.
* Active uncontrolled infection.
* Unstable peptic ulcer, unstable diabetes mellitus or other contraindication for the use of Corticosteroids.
* Inability to take and/or absorb oral medicine
* Prior treatment with capecitabine and/or cisplatin
* Concurrent treatment with other experimental drugs, or participation in another clinical trial with any investigational drug within 30 days prior to study entry

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-11; Primary Completion 2015-10 (Estimated); Study Completion 2016-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Binghe XU, MD, PHD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, ChineseAMS, Beijing, Beijing Municipality, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Cisplatin/Capecitabine: Capecitabine 1000mg/m2 orally Bid on day 1 to day 14 plus Cisplatin 75mg/m2 on day1 of each 21 day cycle, until progression or untolerable toxicity.
  This is a single arm phase II clinical trial.
  Cisplatin/Capecitabine: Cisplatin/Capecitabine: Capecitabine 1000mg/m2 orally Bid on day 1 to day 14 plus Cisplatin 75mg/m2 on day1 of each 21 day cycle, until progression or untolerable toxicity
Period: Overall Study
Arm/Group | Cisplatin/Capecitabine
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cisplatin/Capecitabine
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0
Region of Enrollment [Number; unit: participants]
  China | 33

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Time Frame: 6 months
Measure: Number; unit: percentage of response
Arm/Group | Cisplatin/Capecitabine
Number analyzed (Participants) | 33
percentage of response | 63.6

2. Secondary Outcome: Progression Free Survival
Time Frame: 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Overall Survival
Time Frame: 3 years
Reporting Status: Not Posted

4. Secondary Outcome: Number and Severity of Adverse Events of Patients Enrolled in This Trial
Description: Number and severity of adverse events sufferred by patients who received capecitabine and cisplatin regimen.
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1year
Arm/Group | Cisplatin/Capecitabine
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 27/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin/Capecitabine (N=33)
leukopenia (Blood and lymphatic system disorders) | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes